CLINICAL TRIAL: NCT02436070
Title: Use of Text Messages to Improve Care For Children Following an ED Visit for Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1409-082
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Asthma
Keywords: Pediatrics; Emergency Medicine; Text messaging
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Subjects receive general, health-related text messages applicable for children with asthma.
  Interventions: Behavioral: General text messages
- Test group (Experimental): Subjects receive specific, targeted text messages for post-emergency department discharge asthma care.
  Interventions: Behavioral: Targeted text messages

INTERVENTIONS:
Behavioral: Targeted text messages — Subjects received text messages specific to post ED asthma follow-up
  Arms: Test group
Behavioral: General text messages — Subjects received text messages generalized to children with asthma
  Arms: Control

SUMMARY:
BACKGROUND Asthma is a prevalent and troublesome pediatric condition. In 2013, Emergency Department (ED) providers treated over 3,500 cases of asthma-related complaints at Children's Hospitals and Clinics of Minnesota. Pediatric ED visits for asthma exceeds billions of dollars annually when including direct cost and lost productivity. Many of these visits and resultant costs are avoidable. Patients with well-controlled asthma do not typically exhibit these patterns, while patients with poorly controlled asthma show patterns of increased utilization of healthcare resources and lower quality of life. Evidence suggests that a text message reminder and educational program might positively influence pediatric asthma care practices.

RESEARCH QUESTION Does a targeted ED based text message intervention program improve outpatient follow-up and routine preventive care in pediatric asthma patients?

METHODS Study subjects will be block randomized based on age and insurance group. The experimental group will receive text messages with guidance towards follow-up care with their PCP and the importance of the flu vaccine for children with asthma. The control group will receive a series of educational self-care and health based text messages unrelated to asthma or the flu vaccine. Some self-report of behaviors will be captured via text message response.

ANALYSIS Primary outcomes for the educational versus targeted text message groups will be compared use Chi-square tests. Additional adjustments may be applied for missing data or if, despite randomization, there is substantial imbalance between group in key covariates (eg race/ethnicity, insurance type or asthma severity.)

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of patients aged 4 - 17 years (inclusive) will be eligible for study participation if they meet the following criteria:

  1. Presentation to the ED with a chief complaint related to an asthma exacerbation such as shortness of breath, respiratory distress, wheezing, etc…
  2. Receive an albuterol treatment in the ED
  3. Previous history of asthma as represented in the medical record or by parental report
  4. Have a cell phone that is able to receive text messages
  5. Able to communicate and provide consent in English or Spanish

Exclusion Criteria:

* Caregivers of patients will be excluded from this study for the following reasons:

  1. First episode of wheezing
  2. Admitted to the hospital
  3. Co-morbid respiratory disease:

     1. Cystic fibrosis
     2. Bronchiectasis
     3. Pulmonary hypertension
     4. Other chronic lung disease
  4. Current cancer diagnosis
  5. Previous cardiovascular surgery
  6. Inflammatory bowel disease
  7. Sickle Cell disease

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Follow-up care with primary care provider | 1 week after emergency department discharge
  Assessed via text and follow-up call if no response to text message

SECONDARY OUTCOMES:
Influenza vaccine | 30 days after emergency department discharge
  Assessed via text and follow-up call if no response to text message
Return visit to the emergency department | 30 days after the inaugural emergency department visit
  Assessed via text and follow-up call if no response to text message; Our health record also checked for return visits

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospitals and Clinics of Minnesota - Emergency Department, Minneapolis, Minnesota
  - Children's Minnesota, Saint Paul, Minnesota